CLINICAL TRIAL: NCT05699720
Title: Effect of Nebulized Magnesium Sulphate in Terms of In-hospital Outcome of Patients Admitted With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Acute Exacerbation of COPD and Nebulized Magnesium Sulphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fawad Ahmad Randhawa, Associate Professor, King Edward Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7372/REG/KEMU2018
Record Dates: First submitted 2021-12-15; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulphate (Experimental): Conventional treatment and 250mg of MgSO4 through nebulizer four times a day. 1 vial of injection MgSO4 was taken which contains 1gm of MgSO4 (each vial contains 10ml). It was divided into 4 equal parts, each contained 250mg MgSO4 i.e., 2.5 ml solution, which were used for nebulization 4 times a day.
  Interventions: Drug: Nebulized Magnesium Sulphate
- Conventional (No Intervention): conventional treatment in the form of oxygen inhalation, anti-cholinergic and beta-2 agonist nebulization, intravenous steroids, as well as intravenous antibiotics.

INTERVENTIONS:
Drug: Nebulized Magnesium Sulphate — Group A received 250mg of MgSO4 /dose given through nebulizer four times a day, while group B did not. The groups will be followed for five days to see the results in terms of in-hospital outcome, whether the patient is discharged after fulfilling the set criteria or needing assisted ventilation.
  Arms: Magnesium Sulphate

SUMMARY:
This study is designed to determine the effect of Nebulized Magnesium Sulphate as an add-on therapy with conventional treatment on In-hospital outcome in patients having acute exacerbation of COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is called as the second highly common respiratory disorder after pulmonary Tuberculosis in Pakistan. It is characterized by chronic and progressive breathlessness, cough, sputum production and airflow obstruction, which progressively lead to restricted activity and impaired life quality (1). According to the World Health Organization, COPD would be the third leading cause of mortality by 2020. It imposes a significant economic burden on account of its morbidity (2). This chronic debilitating disorder is accompanied by various comorbid factors that contribute to a spiral of decline, leading to an increase in mortality (3). Episodes of acute deterioration associated with COPD is called exacerbations. These exacerbations are among one of the most common causes of hospital admissions in the country. Acute exacerbation is triggered by bacterial and viral infections and can also be precipitated by environmental factors, including air pollution, second-hand smoke, and periodically variations, i.e., low temperature (winter season) (1). Acute exacerbation lead to deterioration in the patients' quality of life, adverse effects on symptoms and lung functions that may last for many weeks, reduction in lung functions, frequent hospital visits, increase in health expenditure, and significant mortality as lung function cannot recover entirely afterwards (1,2). Acute exacerbations of COPD are treated by oxygen, inhaled bronchodilators, i.e., beta-2 agonists and anticholinergics, antibiotics, and steroids (2,3).

Exacerbations, during the illness, drastically affect the quality of life of the patient, put a burden on healthcare expenses, and are associated with an increase in mortality. Exacerbations also result in the worsening of airway obstruction and an increase in the inflammatory response (5). While smoking is said to be the most significant risk factor in the etiology of COPD, infections mainly account for recurrent episodes of exacerbation occurring during this illness. With advancing industrialization, environmental factors in the form of increasing air pollution contribute to COPD exacerbation pathogenesis (1,2). Effective management of acute exacerbations of COPD will slow disease progression, improve the patient's health status, and lessen the burden on healthcare services (5). It increases interest in optimizing COPD treatment and devising new modalities to prevent episodes of exacerbations. Pulmonary rehabilitation, oxygen inhalation, inhaled and systemic corticosteroids, bronchodilators (β2-agonists and anticholinergic agents), and, if required, mechanical ventilation constitute the standard treatment regimen in COPD. There is a compelling interest in devising increased new strategies to effectively manage and decrease the severity and frequency of exacerbations (4).

Magnesium is a Calcium-mediated bronchodilator that acts with different mechanisms such as calcium antagonism via Calcium-Channels and counteraction of Calcium-medicated smooth muscle contraction, inhibiting the release of Histamine and Acetylcholine from mast cells and cholinergic nerve endings, respectively (2). It is proven that Magnesium helps in providing enhanced bronchodilator effect in acute exacerbations of asthma. However, fewer data and conflicting results are seen regarding its use in acute aggravation of COPD. So far, only six studies have investigated the bronchodilator efficacy of magnesium sulphate in COPD. Intravenous administration of Magnesium during exacerbations of chronic obstructive pulmonary disease (COPD) resulted in the improvement of peak flow.

Randomized, single-blinded, placebo-controlled trials showed that intravenous magnesium sulphate (MgSO4), when given as an adjunct to standard therapy in severe acute asthma, causes pulmonary function improvement and decreases in-hospital admissions (4). Nebulized MgSO4, either separately or in combination with salbutamol, has a visible bronchodilator impact in severe asthma and shows proven betterment (5).

Acute intravenous magnesium in stable COPD patients resulted in a decline of lung hyperinflation as well as improved respiratory muscle strength (5). There are very few placebo-based clinical trials evaluating the efficacy of magnesium sulphate administered via intravenous, nebulized, or both routes in COPD exacerbations. One such trial showed that Intravenous administration of magnesium sulphate has no bronchodilating effect in patients with COPD exacerbations. However, it enhances the bronchodilating effect of other inhaled short-acting bronchodilators (6). Nebulized magnesium sulphate, when added to standard bronchodilator treatment, provides additional relief of dyspnea in patients of acute exacerbations (2). However, these studies showed inconclusive results, and the clinical potential of Magnesium deserves to be further investigated.

Nebulized magnesium sulphate may show promising bronchodilator effect as an add-on therapy to the conventional treatment for COPD exacerbations due to its intracellular effects. In case of a positive outcome, this practice can be incorporated in the management of COPD in its acute exacerbations because of its low cost, being readily available in our hospital settings, convenient mode of administration, and lesser side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. The age of patient should between 30 to 70 years. 2. The patient could be male or female. 3. The duration of COPD must be less than 10 years. 4. Acute exacerbation of COPD requiring hospital admission and any two out of four criteria: I. Increase in the purulence or quantity of sputum II. Dyspnea grade 3, 4 or 5 according to MRC scale (Annexure attached) III. PEFR <200 L/min IV. Respiratory acidosis on arterial blood gas analysis

Exclusion Criteria:

- 1. Known case of other pulmonary parenchymal disease diagnosed by history, examination and previous medical records.

2. Bronchogenic carcinoma diagnosed by history and previous records. 3. Pulmonary edema diagnosed based on history, examination and investigations.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
In- Hospital Outcome | 5 days
  discharge or death or clinical improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Fawad Ahmad Randhawa, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No